CLINICAL TRIAL: NCT07168187
Title: The Effect of Reflexology Treatment on Maternal Anxiety During Induction of Labor With an Extra-amniotic Balloon
Brief Title: The Effect of Reflexology on Time to Delivery During Induction of Labor
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0011-25-WOMC
Record Dates: First submitted 2025-06-08; First posted 2025-09-11 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Reflexology; Labor Induction; Extra Amniotic Balloon
Keywords: induction to delivery time; labor induction; maternal anxiety
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reflexology during induction of labor (Experimental): Participants randomized to this arm will receive a reflexology treatment administered by a certified reflexologist. The session will occur shortly after placement of the extra-amniotic balloon (EAB) for labor induction and before the balloon's spontaneous expulsion or removal at 24 hours. Reflexology will be performed on specific pressure points on the feet, following a standardized protocol intended to reduce maternal anxiety and pain. Participants will also receive routine obstetric care as per institutional protocol.
  Interventions: Other: Reflexology
- Standard care (No Intervention): Participants randomized to this arm will receive standard obstetric care for labor induction with an extra-amniotic balloon (EAB) according to the hospital's clinical protocol. No reflexology or sham procedure will be administered. Anxiety and pain assessments will be conducted at comparable time points to those in the intervention group.

INTERVENTIONS:
Other: Reflexology — Reflexology, a complementary therapy rooted in ancient practices, involves applying pressure to specific points on the feet, hands, or ears thought to stimulate nerve pathways, potentially promoting relaxation and reducing stress. Evidence supporting reflexology's role in obstetrics is growing, with studies highlighting its ability to reduce anxiety, alleviate pain, and influence the duration of labor. Moreover, when reflexology was applied during the active phase of labor it was related to a significant reduction in labor pain intensity and improvements in maternal satisfaction.
  Arms: reflexology during induction of labor

SUMMARY:
This prospective, randomized controlled trial evaluates the effect of reflexology on maternal anxiety, labor duration, and pain in women undergoing labor induction with an extra-amniotic balloon (EAB). Eligible participants are women with a singleton, term pregnancy, cephalic presentation, intact membranes, and a Bishop score <6, without prior cesarean delivery or contraindications to vaginal delivery.

Participants will be randomized to two groups: an intervention group receiving reflexology by a certified practitioner following EAB placement, and a control group receiving standard care. Maternal anxiety will be assessed using the State-Trait Anxiety Inventory (STAI) before and after the intervention. Labor duration and pain scores will also be recorded.

The study plans to enroll 84 participants over two years. Reflexology is a safe, non-invasive complementary therapy, and this study aims to determine whether it provides measurable benefits during labor induction.

DETAILED DESCRIPTION:
Labor induction is a common obstetric procedure that can be associated with maternal anxiety, pain, and prolonged labor, potentially affecting the birth experience and maternal well-being. Complementary interventions may help reduce these effects and improve patient satisfaction.

Reflexology is a non-invasive therapy involving targeted pressure on specific points of the feet, hands, or ears, which may promote relaxation and reduce stress and pain. Preliminary evidence suggests reflexology can decrease maternal anxiety and labor pain, but high-quality data in the context of mechanically induced labor are limited.

This study evaluates reflexology during labor induced with an extra-amniotic balloon (EAB). Participants will be randomized to receive either reflexology by a trained practitioner after EAB placement or standard care without reflexology. Maternal anxiety, labor duration, pain, and patient satisfaction will be systematically assessed, using validated measures for anxiety and pain, along with routine clinical and neonatal data collected from hospital records.

The study aims to enroll 84 participants over two years. All participants will provide informed consent, and data will be de-identified to ensure privacy. This trial seeks to provide evidence on the efficacy of reflexology as a complementary intervention during labor induction, informing clinical practice and enhancing maternal-centered care.

ELIGIBILITY:
Inclusion Criteria:

* Age of ≥18 years
* Gestational age of >37 weeks
* Vertex presentation
* Intact membranes
* Station of the fetus's head < S-4
* Bishop score of <6.

Exclusion Criteria:

* Patients who had undergone a previous cesarean delivery
* Patients with a contraindication for vaginal delivery
* Patients with a known fetal malformation patients undergoing termination of pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Maternal anxiety during labor as perceived by the validated state-trait anxiety index | first STAI questionnaire after recruitment and before induction initiation to assess baseline anxiety. Within 2-10 hours of EAB placement she will fill the second STAI form (similar) and delta STAI score will be calculated
  state-trait anxiety index (STAI-S) questionnaire

SECONDARY OUTCOMES:
Time from Extra-Amniotic Balloon (EAB) placement to balloon expulsion | From the time of EAB placement until the time of balloon expulsion, assessed up to 24 hours after placement.
  The time in hours from the documented placement of the extra-amniotic balloon (EAB) to its spontaneous expulsion from the cervix, recorded by clinical staff or self-reported by the patient. This outcome is used to assess progression of cervical ripening during labor induction. Per developmental protocol, all EABs that do not spontaneously expel within 24 hours will be removed by a physician, and this will be recorded.
Time from labor induction to delivery | From the time of EAB placement until the time of delivery, assessed up to 72 hours after induction initiation.
  Time (in hours) from the initiation of labor induction-defined as the time of extra-amniotic balloon (EAB) placement-to the time of delivery (vaginal or cesarean). This outcome will be used to assess the effect of reflexology on the overall duration of labor after induction.
rate of vaginal birth within 24 hours from induction | 24 hours from induction initiation to delivery
  vaginal birth rate within the first 24 hours from induction initiation in both groups
Pain during labor induction as measured by the Visual Analogue Scale (VAS) | Baseline before EAB placement and post-intervention or within 2-10 hours after EAB placement.
  Maternal perception of pain will be assessed using the Visual Analogue Scale (VAS), a 10 cm horizontal line ranging from 0 to 10, where 0 represents "no pain" and 10 represents "worst imaginable pain." Each participant will report her pain level at two time points:
  1. Baseline (prior to reflexology or standard care), and
  2. After the intervention (reflexology group) or within 2-10 hours after EAB placement (control group).
  The primary pain outcome will be the maximal reported VAS score during the induction process.
Mode of delivery | At delivery
  Mode of delivery categorized as spontaneous vaginal delivery, instrumental vaginal delivery, or cesarean section. Data will be obtained from delivery records.
Maternal satisfaction with the labor induction experience | up to 1 hour from intervention and prior to delivery
  Maternal satisfaction will be assessed using a scale ranging from 1 to 5, where 1 indicates "not satisfied at all" and 5 indicates "maximally satisfied." Participants will rate their satisfaction after the intervention (reflexology or standard care) and before delivery. Higher scores indicate greater satisfaction.
Intrapartum fever | During labor, up to delivery
  Occurrence of maternal intrapartum fever, defined as body temperature ≥38.0°C measured during labor.
Manual lysis of placenta | At delivery
  Need for manual lysis of placenta, defined as manual removal of the placenta following delivery.
Neonatal birthweight | At 1 minute and 5 minutes after birth
  Apgar score at 1 and 5 minutes, each ranging from 0 to 10, with higher scores indicating better neonatal condition.
Umbilical cord pH | At birth
  Arterial umbilical cord pH measured immediately after birth.
NICU admission | Immediately after birth, assessed through hospitalization period (up to 28 days)
  Rate of neonates admitted to the Neonatal Intensive Care Unit (NICU).
Respiratory distress syndrome (RDS) | During initial hospitalization (up to 28 days of life)
  Rate of neonatal respiratory distress syndrome as documented in the neonatal medical record.
Neonatal ventilation | During initial hospitalization (up to 28 days)
  Rate of neonates on mechanical or non-invasive ventilation support during the newborn's hospitalization.
Neonatal neurological morbidity | During initial hospitalization (up to 28 days)
  Rate of neonates with diagnosed neurological complications, including seizures or intraventricular hemorrhage (IVH), during neonatal hospitalization.
Neonatal hypoglycemia | Within first 24 hours after birth
  Rate of neonates with documented blood glucose <40 mg/dL within the first 24 hours of life.
Neonatal blood transfusion | During neonatal hospitalization (up to 28 days)
  Rate of neonates requiring blood transfusion during neonatal hospitalization.
Neonatal phototherapy | During neonatal hospitalization (up to 28 days)
  Rate of neonates admitted for phototherapy for hyperbilirubinemia.
Neonatal death | Up to 28 days after birth
  Rate of dead neonates within the first 28 days of life.

IPD SHARING:
Plan to Share IPD: No